CLINICAL TRIAL: NCT01054326
Title: Effects of Supervised Physical Therapy With Early Activation of the Rotator Cuff Versus Home Exercises in Patients After Arthroscopic Subacromial Decompression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Kalmar County Hospital (Other)
Responsible Party: Kajsa Johansson, PT, Med. Dr, Linköpings University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DNR 02-37
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2006-01

CONDITIONS: Subacromial Decompression
Keywords: arthroscopic subacromial decompression; exercise; physical therapy; rotator cuff; shoulder impingement syndrome; Subacromial impingement after arthroscopic subacromial decompression
MeSH Terms: conditions — Motor Activity; Shoulder Impingement Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supervised physical therapy focusing of rotatorcuff exercises (Experimental): Patients did specific exercises supervised by a physical therapists twice a week during two months. Focus was on early activation of rotator cuff and scapula stabilizers following different phases in a rehabilitation program Assessments before surgery,1 week after as well as 1,2,3 and 6 months after surgery.
  Interventions: Other: Exercises
- Home exercises (Active Comparator): Patients did home exercises following a programme during three months. Assessment considering shoulder function and pain was done before surgery, 1w after as well as 1,2,3 and 6 months after surgery,
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises

SUMMARY:
The objective of this study was to evaluate and compare two different post-surgical rehabilitation strategies, Rehabilitation supervised by a physical therapist including exercises with progressive early activation of the rotator cuff versus basic home exercises regarding shoulder function, pain, health related quality of life and return to work after arthroscopic subacromial decompression.

DETAILED DESCRIPTION:
Patients scheduled for surgery (arthroscopic subacromial decompression)and in the age 25-65 were offered to participate in the study. After surgery they were randomized to either Supervised Physical therapy with early activation of the rotator cuff (PT-group) or to home exercises (H-group). Patients in the PT group met the physical therapist twice a week for exercises and in between these visits they did their exercises at home daily. The H-group did home exercises daily. Shoulder function and pain(primary outcomes)and health related quality of life, returning to work(secondary outcomes)were assessed before surgery, one week after(baseline), 1,2,3 and 6 months after surgery by an independent physical therapist.

ELIGIBILITY:
Inclusion Criteria:

* Subacromial impingement verified with Neer impingement test
* At least 6 month duration of pain
* Treated in primary care without satisfactory results for at least three months.
* Typical history and pain location. Scheduled for surgery (subacromial decompression)
* Three of these four tests must be positive:

  * Neer impingement test
  * Hawkins-Kennedy impingement sign Jobe supraspinatus test
  * Painful arc 60-120 degree

Exclusion Criteria:

* Radiological findings of malignancy osteoarthritis, fractures
* Polyarthritis or fibromyalgia
* Pathological hyper laxity
* Lack of communication skills that prevent the use of outcome measurements
* Cervical spine pathology

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-01; Primary Completion 2006-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Shoulder function and pain | before surgery, 1 w (baseline, 1,2,3 and 6 month after surgery

SECONDARY OUTCOMES:
Health related quality of life and returning to work | before surhery and 1 w(baseline)1,2,3 and 6 months after surgery